CLINICAL TRIAL: NCT03897049
Title: A Randomized Controlled Trial of Trans Women Connected: a Mobile App Delivered Sexual Health Promotion Program
Brief Title: Evaluation of the Trans Women Connected Mobile App for Changes in Sexual Health-related Behavior Among Transgender Women
Acronym: TWC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ETR Associates (Other)
Collaborators: dfusion Inc (Industry); Portland State University (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TransWomenConnected; 5R44MD012279 (NIH)
Record Dates: First submitted 2019-03-25; First posted 2019-04-01 (Actual); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2023-12

CONDITIONS: HIV/AIDS; Health Knowledge, Attitudes, Practice; STI
Keywords: Transgender Women; STI; Sexual Health; HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Behavior; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: This is a two arm randomized controlled trial.
  Implementation. After randomization, participants will be granted access to download and install their respective Trans Women Connected mobile apps (intervention or attention control).
Masking Description: Participants are randomly assigned to their condition without being made aware of their assigned condition. Each condition downloads and uses an app so study activities are similar reducing the likelihood participants will be aware of their assigned condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TWC App (Experimental): The intervention is a mobile app delivered sexual health promotion program designed specifically for transgender women. The mobile app includes 42 interactive activities plus resource maps, opportunities for mentoring, and communication forums for connecting with other transgender women.
  Interventions: Behavioral: Trans Women Connected
- General Health App (Active Comparator): An alternate mobile app (TWC COVID only) designed specifically for transgender women. The mobile app includes 7 interactive activities focused on COVID and COVID resources.
  Interventions: Behavioral: General Health App

INTERVENTIONS:
Behavioral: Trans Women Connected — The intervention will address the unique needs of transgender women and the lack of evidence-based, transgender-specific HIV prevention. It is a mobile app delivered sexual health promotion program that engages transgender women through a strengths based approach to HIV prevention and sexual health that uses the power of social networks to identify and encourage protective factors that support the health of transgender women. This approach recognizes the social and structural barriers that transgender women face. In the context of these barriers, which include stigma and discrimination in a number of interconnected spheres, individually-focused behavioral interventions are insufficient. This intervention takes a more comprehensive approach that intentionally targets community strengths and challenges. The mobile app will include more than 30 interactive activities including resource maps, PrEP/PEP content, and communication forums.
  Arms: TWC App
Behavioral: General Health App — The control group will download a mobile app that addresses COVID and provides COVID resources.
  Arms: General Health App

SUMMARY:
The study is a 2-arm cluster randomized controlled trial to be conducted with 450 trans women to assess the effectiveness of the Trans Women Connected mobile app. Those in the treatment arm will be provided with the Trans Women Connected app, to be downloaded to their own device, and asked to use it during a month period. Those in the control arm will be asked to download a general health app and use it during a month period. Participants will complete brief online surveys at baseline, immediately following the app-use period (1-month post baseline), and at 3- and 6-months following baseline. The baseline and follow-up assessments will collect data on demographic characteristics, measures related to our primary and secondary outcomes, and psychosocial measures. The primary outcome measures are self-reported sexually transmitted infection (STI)/HIV testing and sex without a condom, with secondary measures including sexual risk behaviors, health care visits, perceived social support/connectedness, pre-exposure prophylaxis (PrEP) use, self-efficacy in negotiation/communication, and comfort with gender identity and appearance. In addition, process data, such as forum content, and usage data will be collected and analyzed.

DETAILED DESCRIPTION:
A 2-arm cluster randomized controlled trial will be conducted with 450 trans women to assess the effectiveness of the Trans Women Connected mobile app. The Trans Women Connected intervention will address the unique needs of transgender women and the lack of evidence-based, transgender-specific HIV prevention. It is a mobile app delivered sexual health promotion program that engages transgender women through a strengths-based approach to HIV prevention and sexual health that uses the power of social networks to identify and encourage protective factors that support the health of transgender women. This approach recognizes the social and structural barriers that transgender women face. In the context of these barriers, which include stigma and discrimination in a number of interconnected spheres, individually-focused behavioral interventions are insufficient. This intervention takes a more comprehensive approach that intentionally targets community strengths and challenges. The mobile app will include more than 30 interactive activities including resource maps, PrEP content, post-exposure prophylaxis (PEP) content, and communication forums.

To be eligible, participants will be required to self-identify as transgender women; report having had 2 or more sexual partners in the past 90 days with at least one of those partners having a penis; be age 18-49 at baseline; own a smartphone; and reside in any state in the United States. Those in the treatment arm will be provided with the Trans Women Connected app, to be downloaded to their own device, and asked to use it during a month period. Those in the control arm will be asked to download a general health app and use it during a month period. Participants will complete brief online surveys at baseline, immediately following the app-use period (1-month post baseline), and at 3- and 6-months following baseline.

Participants will be recruited using a variety of methods, including: 1) Regional transwomen recruitment/retention specialists who are responsible for facilitating recruitment in their regions, addressing study questions, and maintaining connections with each participant to support study engagement; 2) Organizations. Organizations from across the U.S., at least one per state, that serve transgender women will be approached to help recruit participants through social media and in-person. 3) Google Adwords. Placing study advertisements on Google based on keyword for participant recruitment has been shown to be effective. 4) Social Media Advertising including targeted advertising on social media sites (Facebook/Instagram) and sponsoring study posts with social media influencers in the Transwomen community. Social media advertising has been shown to be favorable in terms of its cost-effectiveness, usability, and reach, especially with hard-to-reach populations, young adults and lesbian, gay, bisexual, and transgender (LGBT) populations. 5) Participant Recruitment (participants sharing information about the study within their networks). Participants will complete 4 web-based surveys and will receive $20 for baseline survey, $20 for an immediate posttest, $40 at 3-month follow up, $60 at final 6-month follow up.

Randomization. The 2-arm randomized controlled trial involves randomizing individual participants using an equal allocation (allocation ratio 1:1) to receive the full TWC app or an attention control app. Participants were randomized after completing their baseline surveys using the randomizer feature of Qualtrics.

Data Collection. Participants will be surveyed at 4 time points. 1) before randomization, 2) after using the mobile app for 1 month, 3) three months after completion of the baseline, and 4) six months after completion of the baseline. Surveys will be completed online through emailed or texted links. Data will also be collected through the apps. This includes usage data, such as what activities participants used and for how long, and process data, which includes content on the communication forum, text answers in the app, and visual content such as vision boards. Participants will receive an incentive of $20 for the baseline and immediate post-intervention survey, $40 for the 3-month follow up survey, and $60 for the 6 month follow up survey.

Study Hypotheses. Primary Hypotheses 1 (representing sexual health risk reduction through engagement in care 1) Women in the intervention group will report more STI testing (higher rates of STI testing in the prior 90 days) than the comparison group. Primary Hypotheses 2, women in the intervention group will report fewer acts of receptive condomless anal intercourse or condomless vaginal intercourse. Secondary Hypotheses (representing other important sexual health risk, and psychosocial outcomes):1) Participants in the intervention group will report reduced sexual risk taking including fewer acts of receptive condomless anal intercourse or condomless vaginal intercourse; greater use of condom use at last intercourse (receptive anal or vaginal); and increased use of PrEP for those that are HIV- 2) Participants in the intervention group will engage more with proactive health care and report more health care visits. 3) Participants in the treatment group will report more connectedness with other transgender women, including perceived social support and engagement with a mentor. 4) Participants in the intervention group will report greater efficacy in having safer sex and in communication both with partners and health care workers. 5) Those in the treatment group will have greater acceptance of their gender identity/comfort with gender identity.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-49 at the start of the study.
2. self-identify as transgender women
3. self-identify as sexually active with more than one partner in the prior 90 days
4. at least one sexual partner in the last 90 days had a penis
5. has a smartphone
6. resides in the U.S.

Exclusion Criteria:

Anyone not meeting inclusion criteria

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All participants must identify as transgender women.
Enrollment: 574 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Kuhn, Principal Investigator — dfusion Inc
Locations (1):
- ETR, Scotts Valley, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramirez-Valles J, Heckathorn DD, Vazquez R, Diaz RM, Campbell RT. From networks to populations: the development and application of respondent-driven sampling among IDUs and Latino gay men. AIDS Behav. 2005 Dec;9(4):387-402. doi: 10.1007/s10461-005-9012-3. PMID 16235135

RESULTS

PARTICIPANT FLOW:
Groups:
- General Health App: An alternate mobile app (TWC COVID only) was designed specifically for transgender women. The mobile app includes 7 interactive activities focused on COVID and COVID resources.
Period: Overall Study
Arm/Group | TWC App | General Health App
Started | 275 | 299
Completed 1st Follow-up | 182 | 205
Completed 2nd Follow-up | 173 | 191
Completed (Participants are marked as completed if they completed the third follow-up) | 177 | 199
Not Completed | 98 | 100

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TWC App | General Health App | Total
Number analyzed (Participants) | 275 | 299 | 574
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 5 participants did not report age at baseline. 4 control participants and 1 treatment participant.
  years
    number analyzed (Participants) | 274 | 295 | 569
    (all) | 31.59 (7.85) | 31.49 (7.88) | 31.54 (7.86)
Sex/Gender, Customized [Number; unit: participants]
  Transgender woman | 275 | 299 | 574
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 72 | 78 | 150
  Not Hispanic or Latino | 202 | 221 | 423
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 12 | 19
  Asian | 3 | 13 | 16
  Native Hawaiian or Other Pacific Islander | 6 | 8 | 14
  Black or African American | 76 | 90 | 166
  White | 125 | 117 | 242
  More than one race | 39 | 37 | 76
  Unknown or Not Reported | 19 | 22 | 41
Region of Enrollment [Number; unit: participants]
  United States | 275 | 299 | 574
Sexual orientation [Count of Participants; unit: Participants]
  Heterosexual | 69 | 78 | 147
  Not heterosexual | 206 | 221 | 427
STI test in past 3 months [Count of Participants; unit: Participants]
  Tested for STI in past 3 months | 159 | 180 | 339
  Not tested for STI in past 3 months | 106 | 108 | 214
  Not reported | 10 | 11 | 21
HIV test in past 3 months [Count of Participants; unit: Participants]
  Tested for HIV in past 3 months | 137 | 148 | 285
  Not tested for HIV in past 3 months | 75 | 83 | 158
  Not reported | 63 | 68 | 131
Receptive sex without condom in past 3 months [Count of Participants; unit: Participants]
  Had receptive sex without a condom in past 3 months | 208 | 232 | 440
  Did not have receptive sex without a condom in past 3 months | 59 | 57 | 116
  Not reported | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Self-reported HIV or STI Testing in Past 3 Months
Description: Participant reported having tested for HIV or STI in the past 3 months
Time Frame: 3-months post intervention
Population: All participants with baseline and 3-month follow-up survey.
Measure: Count of Participants; unit: Participants
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 98 | 109
Participants | 76 | 88
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.914, Regression, Logistic; Odds Ratio (OR) = 0.961, 95% CI 2-sided [0.463 to 1.994]

2. Primary Outcome: Self-reported HIV or STI Testing in Past 3 Months
Description: Participant reported having tested for HIV or STI in the past 3 months
Time Frame: 6-months post intervention
Population: All participants who completed baseline and 6-month follow-up surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 95 | 108
Participants | 77 | 88
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.990, Regression, Logistic; Odds Ratio (OR) = 0.979, 95% CI 2-sided [0.473 to 2.074]

3. Primary Outcome: Receptive Condomless Anal Intercourse or Condomless Vaginal Intercourse in Past 3 Months
Description: Participant reported having had receptive anal intercourse without a condom or receptive vaginal intercourse without a condom in the past 3 months
Time Frame: 3-months post intervention
Population: All participants who completed baseline and 3-month follow-up surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 154 | 165
Participants | 106 | 101
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.167, Regression, Logistic; Odds Ratio (OR) = 1.434, 95% CI 2-sided [0.861 to 2.390]

4. Primary Outcome: Receptive Condomless Anal Intercourse or Condomless Vaginal Intercourse in Past 3 Months
Description: as for outcome 3
Time Frame: 6-months post intervention
Population: All participants completing baseline and 6-month follow up survey.
Measure: Count of Participants; unit: Participants
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 158 | 168
Participants | 99 | 96
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.118, Regression, Logistic; Odds Ratio (OR) = 1.492, 95% CI 2-sided [0.903 to 2.466]

5. Secondary Outcome: Use of a Condom at Last Receptive Anal Intercourse or Vaginal Intercourse
Description: Participant reported using a condom at last receptive anal intercourse or vaginal intercourse
Time Frame: 3-month post intervention
Population: All participants who completed baseline and 3-month follow-up surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 171 | 164
Participants | 55 | 51
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.265, Regression, Logistic; Odds Ratio (OR) = 1.335, 95% CI 2-sided [0.803 to 2.221]

6. Secondary Outcome: Use of a Condom at Last Receptive Anal Intercourse or Vaginal Intercourse
Description: Participant reported using a condom at last receptive anal intercourse or vaginal intercourse
Time Frame: 6-month post intervention
Population: All participants who completed baseline and 6-month follow-up surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 167 | 181
Participants | 48 | 52
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.971, Regression, Logistic; Odds Ratio (OR) = 0.990, 95% CI 2-sided [0.593 to 1.654]

7. Secondary Outcome: Health Care Visits in Past 3 Months
Description: Average # of self-reported visits to a health care provider (of any type and by type)
Time Frame: 3-months post intervention
Population: All participants completing baseline and 3-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 167 | 178
Number of visits | 4.75 (5.49) | 5.02 (4.94)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.942, Regression, Linear; Mean Difference (Net) = -0.27

8. Secondary Outcome: Health Care Visits in Past 3 Months
Description: Average # of self-reported visits to a health care provider (of any type and by type)
Time Frame: 6-months post intervention
Population: All participants completing baseline and 6-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 169 | 191
Number of visits | 4.63 (4.54) | 4.61 (4.10)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.741, Regression, Linear; Mean Difference (Net) = 0.02

9. Secondary Outcome: Mini-Medical Outcomes Study--Social Support Survey (mMOS-SS)
Description: Perceptions of social support, mean score of 8 items measured on a five point scale (1-5). Scale range is from 1 - 5 with a higher number indicating greater perceived social support, which is a better outcome.
Time Frame: 1-month post intervention
Population: All participants completing baseline and 1-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 173 | 185
score on a scale | 3.23 (1.18) | 3.16 (1.08)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.494, Regression, Linear; Mean Difference (Net) = 0.07

10. Secondary Outcome: Mini-Medical Outcomes Study--Social Support Survey (mMOS-SS)
Description: as for outcome 9
Time Frame: 3-month post intervention
Population: All participants completing baseline and 3-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 168 | 176
score on a scale | 3.30 (1.15) | 3.15 (1.16)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.651, Regression, Linear; Mean Difference (Net) = 0.15

11. Secondary Outcome: Mini-Medical Outcomes Study--Social Support Survey (mMOS-SS)
Description: as for outcome 9
Time Frame: 6-month post intervention
Population: All participants completing baseline and 6-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 168 | 185
score on a scale | 3.46 (1.14) | 3.16 (1.09)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.022, Regression, Linear; Mean Difference (Net) = 0.30

12. Secondary Outcome: Engaged as/With Mentor in Past 3 Months
Description: Self-reported number of contacts in the past 3 months as a mentor/mentee for guidance or support
Time Frame: 3-months post intervention
Population: Participants completing baseline and 3-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: Number of mentee/mentor contacts
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 20 | 12
Number of mentee/mentor contacts | 5.35 (8.53) | 2.50 (1.00)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.189, Regression, Linear; Mean Difference (Net) = 2.85

13. Secondary Outcome: Engaged as/With Mentor in Past 3 Months
Description: Self-reported number of contacts, in the past 3 months, as a mentor/mentee for guidance or support
Time Frame: 6-months post intervention
Population: Participants completing baseline and 6-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: Number of mentor/mentee contacts
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 19 | 12
Number of mentor/mentee contacts | 6.32 (10.00) | 3.25 (1.55)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.218, Regression, Linear; Mean Difference (Final Values) = 3.07

14. Secondary Outcome: PrEP Uptake
Description: Self-reported uptake of PrEP among HIV since last measurement period- subsample
Time Frame: 1-month post intervention
Population: Participants completing baseline and 1-month follow-up survey.
Measure: Count of Participants; unit: Participants
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 126 | 141
Participants | 6 | 13
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.149, Regression, Logistic; Odds Ratio (OR) = 0.479, 95% CI 2-sided [0.173 to 1.305]

15. Secondary Outcome: PrEP Uptake
Description: Self-reported uptake of PrEP among HIV since last measurement period- subsample
Time Frame: 3-month post intervention
Population: Participants completing baseline and 3-month follow-up surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 107 | 119
Participants | 8 | 8
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.839, Regression, Logistic; Odds Ratio (OR) = 1.111, 95% CI 2-sided [0.403 to 3.063]

16. Secondary Outcome: PrEP Uptake
Description: Self-reported uptake of PrEP among HIV since last measurement period- subsample
Time Frame: 6-month post intervention
Population: Participants completing baseline and 6-month follow-up survey.
Measure: Count of Participants; unit: Participants
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 96 | 128
Participants | 8 | 4
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.063, Regression, Logistic; Odds Ratio (OR) = 3.302, 95% CI 2-sided [0.937 to 11.641]

17. Secondary Outcome: Condom/Barrier Negotiation Self Efficacy Scale
Description: Scale measures self-efficacy in decisions around using protective barriers during sex. Average of 8 items on a 7-point scale (1 to 7), with a range of 1 - 7, with a higher score indicating better outcomes, or greater self-efficacy
Time Frame: 1 month post-intervention
Population: Participants completing baseline and 1-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 177 | 188
score on a scale | 5.40 (1.58) | 5.48 (1.59)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.650, Regression, Linear; Mean Difference (Net) = -0.08

18. Secondary Outcome: Condom/Barrier Negotiation Self Efficacy Scale
Description: as for outcome 17
Time Frame: 3- month post intervention
Population: Participants completing baseline and 3-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 170 | 179
score on a scale | 5.63 (1.51) | 5.54 (1.49)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.531, Regression, Linear; Mean Difference (Net) = 0.09

19. Secondary Outcome: Condom/Barrier Negotiation Self Efficacy Scale
Description: as for outcome 17
Time Frame: 6-month post intervention
Population: Participants completing baseline and 6-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 171 | 189
score on a scale | 5.52 (1.60) | 5.55 (1.54)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.761, Regression, Linear; Mean Difference (Net) = -0.03

20. Secondary Outcome: Health Education Impact Questionnaire (heiQ) Health Services Navigation Sub-Scale
Description: Sub-scale measures comfort navigating health services. Average of 5 items on a 4-point scale (1-4), with a range of 1 - 4, with a higher score indicating greater comfort navigating health services
Time Frame: 1-month post intervention
Population: Participants completing baseline and 1-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 174 | 185
score on a scale | 3.14 (0.86) | 3.03 (0.86)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.503, Regression, Linear; Mean Difference (Net) = 0.11

21. Secondary Outcome: Health Education Impact Questionnaire (heiQ) Health Services Navigation Sub-Scale
Description: as for outcome 20
Time Frame: 3-month post intervention
Population: Participants completing baseline and 3-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 169 | 184
score on a scale | 3.17 (0.88) | 3.16 (0.80)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.541, Regression, Linear; Mean Difference (Net) = 0.01

22. Secondary Outcome: Health Education Impact Questionnaire (heiQ) Health Services Navigation Sub-Scale
Description: as for outcome 20
Time Frame: 6- month post intervention
Population: Participants completing baseline and 6-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 168 | 183
score on a scale | 3.18 (0.88) | 3.20 (0.77)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.537, Regression, Linear; Mean Difference (Net) = -0.02

23. Secondary Outcome: Transgender Congruence Scale (TCS)
Description: Scale measures degree of comfort with external appearance as it relates to gender identity. Average of 12 items on a 5-point scale, with a range of 1 - 5, with a higher score indicating a perception that their appearance reflects their chosen gender identity
Time Frame: 1-month post intervention
Population: Participants completing baseline and 1-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 174 | 184
score on a scale | 3.65 (0.94) | 3.46 (0.91)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.057, Regression, Linear; Mean Difference (Net) = 0.19

24. Secondary Outcome: Transgender Congruence Scale (TCS)
Description: as for outcome 23
Time Frame: 3-month post intervention
Population: Participants completing baseline and 3-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 166 | 178
score on a scale | 3.61 (0.93) | 3.51 (0.95)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.402, Regression, Linear; Mean Difference (Net) = 0.10

25. Secondary Outcome: Transgender Congruence Scale (TCS)
Description: as for outcome 23
Time Frame: 6-month post intervention
Population: Participants completing baseline and 6-month follow-up surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 164 | 187
score on a scale | 3.66 (0.90) | 3.51 (0.92)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.308, Regression, Linear; Mean Difference (Net) = 0.15

26. Secondary Outcome: Trans Women Connected Satisfaction Survey
Description: Scale measures participants' reactions to the app. Average of 3 items on a 5-point scale with a range of 1 to 5 with a higher score indicating greater levels of satisfaction with the app.
Time Frame: 1-month post intervention
Population: Participants completing 1-month follow-up survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TWC App | General Health App
Number analyzed (Participants) | 150 | 166
score on a scale | 4.06 (0.96) | 3.58 (1.20)
Statistical Analysis 1: Comparison: TWC App vs General Health App; Test type: Superiority; p = 0.001, Regression, Linear; Mean Difference (Net) = 0.48

ADVERSE EVENTS:
Time Frame: Entire study period (consent through 6 month follow-up), approximately 7 months.
Description: Used "clinicaltrials.gov" definitions.
Arm/Group | TWC App | General Health App
All-Cause Mortality (participants affected / at risk) | 0/275 | 0/299
Serious Adverse Events (participants affected / at risk) | 0/275 | 0/299
Other Adverse Events (participants affected / at risk) | 0/275 | 0/299

LIMITATIONS AND CAVEATS:
Relatively brief follow-up period (6 months) limits insights on longer-term impacts; some participants reported struggles with app download (affected both conditions), which may be linked to lack of more robust treatment effects; COVID impacted study progression and likely impacted behavior related to some outcomes (e.g., HIV/STI testing due to service shifts affected by COVID).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT03897049/Prot_SAP_000.pdf